CLINICAL TRIAL: NCT07275346
Title: Evaluating Surgical Approaches for Medium-to-Large Ventral Hernias: Open, Laparoscopic, and Robotic-Assisted Techniques
Brief Title: Surgical Approaches for Medium-to-Large Ventral Hernias: Open, Laparoscopic, and Robotic-Assisted Techniques
Status: Active, not recruiting | Type: Observational
Sponsor: Andreas Älgå (Other)
Collaborators: Danderyds Hospital, Stockholm, Sweden (Unknown); Sodertalje Hospital (Other); Ersta Hospital, Sweden (Other); Stockholm South General Hospital (Other)
Responsible Party: Sponsor-Investigator, Andreas Älgå, Principal Investigator, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Other Study IDs: VH-OpenLapRob
Record Dates: First submitted 2025-11-19; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Ventral Hernia
Keywords: laparoscopic surgery; robot-assisted surgery; ventral hernia; surgery
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Open surgery: Patents who had open surgery for their ventral hernia
- Conventional laparoscopic surgery: Patents who had conventional laparoscopic surgery for their ventral hernia
- Robot-assisted laparoscopic surgery: Patents who had robot-assisted laparoscopic surgery for their ventral hernia

SUMMARY:
The purpose of this project is to investigate whether the use of the new robot-assisted technique in surgery for large and medium-sized ventral midline hernias has brought tangible benefits to patients in terms of Textbook outcome, length of stay, complications and recurrence, compared to open technique and conventional laparoscopic technique. In addition, the investigators will assess the health economic aspects of the different techniques.

DETAILED DESCRIPTION:
In the Stockholm Region, ventral hernia surgeries are performed at Södersjukhuset, Danderyds Hospital, Södertälje Hospital, Norrtälje Hospital, St Göran Hospital, Ersta Hospital and Karolinska Hospital. The hospitals differ in terms of admission areas, profile areas and access to surgical robots for hernia surgery. Since the introduction of robot-assisted surgery in Stockholm around 2017-2018, Södersjukhuset and Danderyd Hospital have used this technology to varying extents for ventral hernia, while the other hospitals have only offered open and conventional laparoscopic surgery. There is no established distribution of hernia patients in the region and no joint treatment conferences. The patients have therefore been distributed primarily depending on place of residence and referral patterns between the hospitals, which has also influenced the choice of method. Similar hernia patients have thus been offered different surgical treatments depending on which hospital in Stockholm the patient was treated at.

The robotic platform involves significant investment costs and costs for robotic instruments. Several studies also indicate that the surgical time is often longer, which can also increase costs. However, the promising results with shorter hospital stay and fewer complications could outweigh the increased surgical costs that have been demonstrated in several studies. The investigators will compare the costs of robot-assisted ventral hernia surgery in the operating room, in the hospital and after discharge with the corresponding costs for open and conventional laparoscopic surgery. Cost-effectiveness analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Large and medium-sized midline hernias (EHS classification W2-W3)

Exclusion Criteria:

* Hernia operations combined with bowel procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients registered in the Swedish Abdominal Hernia Registry and operated on at Södersjukhuset, Ersta Hospital, Danderyd Hospital, or Södertälje Hospital
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
% of patients with Textbook Outcome | 1 month post surgery
  Textbook Outcome is a composite outcome that will be used as a measure of a problem-free postoperative recovery. Textbook Oitcome will be defined as the absence of complications, prolonged hospital stay, readmission, and reoperation. Textbook Outcome is a binary outcome measure; the patient will either have Textbook Outcome (i.e. a problem-free postoperative recovery) or not (i.e. not a problem-free postoperative recovery).

SECONDARY OUTCOMES:
Rate of.post operative complications | 1 month post surgery
  Post operative complications defined as Clavien-Dindo grade III or higher
Recurrence | 2-7 years post surgery
  A recurrence of the patients ventral hernia. Re-operation will be used as a proxy for recurrence.
Length of stay | Perioperatively
  Length of hospital stay for the surgery
Cost | Up to 1 year post surgery
  The costs of the three different surgical methods for ventral hernias. Cost-effectiveness calculations will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Älgå, MD, PhD, Principal Investigator — Karolinsk Institutet
Locations (1):
- Karolinska Institutet, Södersjukhuset, Stockholm, Sweden